CLINICAL TRIAL: NCT02969798
Title: Preservation of Beta Cell Function in Pre-diabetes in Subject With Impaired Fasting Glucose (IFG) and Impaired Glucose Tolerance (IGT)
Brief Title: Pre-diabetes in Subject With Impaired Fasting Glucose (IFG) and Impaired Glucose Tolerance (IGT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American Diabetes Association (Other); AstraZeneca (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20130414H; R01DK024092-34 (NIH)
Record Dates: First submitted 2016-03-16; First posted 2016-11-21 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Impaired Glucose Tolerance (IGT); Impaired Fasting Glucose (IFG)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — dapagliflozin; saxagliptin; Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Healthy normal glucose tolerance (NGT) subjects (No Intervention): Subjects (Fasting Plasma Glucose or FPG < 100 mg/dl and 2-h PG < 140 mg/dl) without FH (family history) of diabetes in a first degree relative
- Isolated IGT with Dapagliflozin (Active Comparator): Healthy subjects with isolated IGT (FPG < 100; 2-h PG = 140-199) will receive dapagliflozin, 10 mg/day
  Interventions: Drug: Dapagliflozin
- Isolated IGT with Saxagliptin (Active Comparator): Healthy subjects with isolated IGT (FPG < 100; 2-h PG = 140-199) will receive saxagliptin, 5 mg/day
  Interventions: Drug: Saxagliptin
- Isolated IGT with Pioglitazone (Active Comparator): Healthy subjects with isolated IGT (FPG < 100; 2-h PG = 140-199) will receive pioglitazone, the dose will increase from 15 mg/day to 30 mg/day at month two
  Interventions: Drug: Pioglitazone
- Isolated IGT with Metformin (Active Comparator): Healthy subjects with isolated IGT (FPG < 100; 2-h PG = 140-199) will receive Metformin, starting at 1000 mg/day and increased to 2000 mg/day at month 2.
  Interventions: Drug: Metformin
- Isolated IFG with Dapagliflozin (Active Comparator): Healthy subjects with isolated IFG (FPG = 100-125; 2-h PG < 140) will receive dapagloflozin, 10mg/day
  Interventions: Drug: Dapagliflozin
- Isolated IFG with Saxagliptin (Active Comparator): Healthy subjects with isolated IFG (FPG = 100-125; 2-h PG < 140) will receive saxagliptin, 10mg/day
  Interventions: Drug: Saxagliptin
- Isolated IFG with Pioglitazone (Active Comparator): Healthy subjects with isolated IFG (FPG = 100-125; 2-h PG < 140) will receive pioglitazone, the dose will increase from 15 mg/day to 30 mg/day at month two
  Interventions: Drug: Pioglitazone
- Isolated IFG with Metformin (Active Comparator): Healthy subjects with isolated IFG (FPG = 100-125; 2-h PG < 140) will receive Metformin, starting at 1000 mg/day and increased to 2000 mg/day at month 2.
  Interventions: Drug: Metformin
- IGT plus IFG with Dapagliflozin (Active Comparator): Healthy subjects with IGT plus IFG will receive dapagliflozin, 10mg/day
  Interventions: Drug: Dapagliflozin
- IGT plus IFG with Saxagliptin (Active Comparator): Healthy subjects with IGT plus IFG will receive saxagliptin, 10mg/day
  Interventions: Drug: Saxagliptin
- IGT plus IFG with Pioglitazone (Active Comparator): Healthy subjects with IGT plus IFG will receive pioglitazone, the dose will increase from 15 mg/day to 30 mg/day at month two
  Interventions: Drug: Pioglitazone
- IGT plus IFG with Metformin (Active Comparator): Healthy subjects with IGT plus IFG will receive Metformin, starting at 1000 mg/day and increased to 2000 mg/day at month 2.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — 10mg/day
  Other Names: farxiga
  Arms: IGT plus IFG with Dapagliflozin; Isolated IFG with Dapagliflozin; Isolated IGT with Dapagliflozin
Drug: Saxagliptin — 5mg/day
  Other Names: onglyza
  Arms: IGT plus IFG with Saxagliptin; Isolated IFG with Saxagliptin; Isolated IGT with Saxagliptin
Drug: Pioglitazone — the dose will increase from 15 mg/day to 30 mg/day at month two
  Other Names: actos
  Arms: IGT plus IFG with Pioglitazone; Isolated IFG with Pioglitazone; Isolated IGT with Pioglitazone
Drug: Metformin — starting at 1000 mg/day and increased to 2000 mg/day at month 2.
  Other Names: glucophage
  Arms: IGT plus IFG with Metformin; Isolated IFG with Metformin; Isolated IGT with Metformin

SUMMARY:
HYPOTHESIS: Impaired glucose tolerance (IGT) and impaired fasting glucose (IFG) have distinct pathophysiologic etiologies. Therefore, therapeutic interventions designed to correct the specific underlying pathogenic abnormalities in IGT and IFG will be required to optimally prevent the progressive beta cell failure and development of overt type 2 diabetes.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

1. To examine the effect of the following pharmacologic interventions on beta cell function, insulin sensitivity, and glucose tolerance status in individuals with isolated impaired glucose tolerance (IGT): (i) treatment with the renal Sodium-glucose co-transporter 2 (SGLT2) inhibitor inhibitor, dapagliflozin; (ii) treatment with the inhibitors of dipeptidyl peptidase 4, also DPP4, saxagliptin ; (iii) treatment with the thiazolidinedione, pioglitazone; (iv) treatment with the biguanide, metformin.
2. To examine the effect of the following pharmacologic interventions on beta cell function, insulin sensitivity, and glucose tolerance status in individuals with isolated impaired fasting glucose (IFG): (i) treatment with the renal SGLT2 inhibitor, dapagliflozin; (ii) treatment with the DPP4 inhibitor, saxagliptin; (iii) treatment with the thiazolidinedione, pioglitazone; (iv) treatment with the biguanide, metformin.
3. To examine the effect of the following pharmacologic interventions on beta cell function, insulin sensitivity, and glucose tolerance status in individuals with combined impaired glucose tolerance (IGT) plus impaired fasting glucose (IFG): i) treatment with the renal SGLT2 inhibitor, dapagliflozin; (ii) treatment with the DPP4 inhibitor, saxagliptin; (iii) treatment with the thiazolidinedione, pioglitazone; (iv) treatment with the biguanide, metformin.

ELIGIBILITY:
Inclusion Criteria:

* NGT subjects will serve as controls and will be matched in age, gender, ethnicity, and BMI to IGT and IFG subjects

  1. Male or female subjects between the ages of 18 and 65 years of age, inclusive, at Screening.
  2. FPG < 100 mg/dl and 2-h PG < 140 mg/dl
  3. BMI = 24-40 kg/m2;
  4. Stable body weight (±4lbs) over the preceding 3 months
  5. Subjects with no evidence of major organ system disease as determined by physical exam, history, and screening laboratory data
  6. Females of childbearing potential with a negative pregnancy test at Screening and Treatment visits, using one of the following forms of contraception for the duration of participation in the study (i.e., until Follow-up 7-14 days post last dose):

     * Oral contraceptive
     * Injectable progesterone
     * Subdermal implant
     * Spermicidal foam/gel/film/cream/suppository
     * Diaphragm with spermicide
     * Copper or hormonal containing IUD
     * Sterile male partner vasectomized > 6 month pre-dosing.
  7. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
  8. Subjects must be willing and able to comply with scheduled visits, treatment, laboratory tests and study procedures.

Exclusion Criteria:

1. Recent (i.e., within three (3) months prior to Screening) evidence or medical history of unstable concurrent disease such as: documented evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, immunological, or clinically significant neurological disease.
2. Subjects with a family history of diabetes in a first degree relative
3. BMI of less than 24 or greater than 40 kg/m2
4. Unstable body weight (change of greater than ±4lbs over the preceding 3 months
5. Subjects participating in an excessively heavy exercise program
6. Subject with a feeding/sleeping schedule different from a daytime feeding/night time sleeping schedule
7. Subjects taking medications known to alter glucose metabolism (with the exception of metformin and/or pioglitazone) or which effect brain neurosynaptic function are excluded.
8. Subjects with evidence of major organ system disease as determined by physical exam, history, and screening laboratory data
9. Pregnant subjects or subjects unwilling to use birth control during their study enrollment
10. Blood donation of approximately 1 pint (500 mL) within 8 weeks prior to Screening.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
12. Subjects with hematuria will be excluded.
13. Subjects with evidence or prior history of heart failure will be excluded
14. Subjects with family history of pancreatic, bladder, and breast cancer will be excluded.
15. Subjects with history of pancreatitis will be excluded.
16. Subjects with eGFR < 60 ±5 ml/min.1.73m2 will be excluded.
17. Subjects with elevated serum creatinine (>1.5 mg/dl males/1.4 mg/dl females) will be excluded.
18. Subjects with a history of orthostatic hypotension (>15/10 mmHg) will be excluded.
19. Subjects with liver enzymes (ALT, AST) >3-fold above upper normal limit will be excluded.
20. Subjects with a history of hypersensitivity to pioglitazone, dapagliflozin, or Saxagliptin will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Beta cell function | 24 months after treatment phase begins
  Beta cell function will be measured as insulin secretion during the hyperglycemic clamp (mean plasma insulin concentration in uU/ml) multiplied by insulin sensitivity measured with the euglycemic insulin clamp (mg/kg.min).
Insulin sensitivity | 24 months after treatment phase begins
  Insulin sensitivity will be measured with the euglycemic insulin clamp and expressed as mg/kg.min.
Glucose tolerance status | 24 months after treatment phase begins
  Glucose tolerance status will be evaluated by measuring the HbA1c which is a measure of the average of the amount of glucose attached to hemoglobin over the past 3 months, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States